CLINICAL TRIAL: NCT03433664
Title: Carbon Dioxide Laser Treatment in Burn-related Scarring: A Prospective Randomised Controlled Trial
Brief Title: Carbon Dioxide Laser Treatment in Burn-related Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Western Australia (Other)
Responsible Party: Principal Investigator, Fiona M. Wood, Head of State Burns Unit WA, The University of Western Australia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/135
Record Dates: First submitted 2018-01-06; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Burns Scarring
Keywords: CO2 laser; Ablative fractional laser
MeSH Terms: interventions — Lasers, Gas

STUDY DESIGN:
Intervention Model Description: Scar area (10x10cm square) randomly assigned a square vector 'map' which split the scar into a control and treatment half along one of 4 vectors: vertical, horizontal, and along both diagonals. The envelope revealing the vector map and treatment zones was opened by the treating laser clinician immediately prior to the first treatment. The same treating clinician performed all laser treatments to minimise inter-user variability.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patient and treating clinician were aware of which scar half had been treated, however investigator and assessor were blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental): Each treatment half of the scar received three standardised CO2 laser treatments using the DeepFX setting hand piece (Ultrapulse, Lumenis), performed under general anaesthetic at 4-6 week intervals. All treatments consisted of a single pass of 300Hz, 5% density and 50mJ energy with minimal overlapping. Post-operatively all laser treatment and control zones had emollient applied and silicone dressings which were removed at 48 hours. Further emollient was applied twice daily for 2 weeks to all areas of the scar. Standard care scar management (including silicone, massage and pressure garments) was directed by burn occupational therapists and was continued for all areas of scar.
  Interventions: Device: CO2 laser
- Control (No Intervention): Each control half of the scar received emollient applied twice daily for 2 weeks to all areas of the scar after each treatment. Standard care scar management (including silicone, massage and pressure garments) was directed by burn occupational therapists and was continued for all areas of scar.

INTERVENTIONS:
Device: CO2 laser — Fractional CO2 laser treatment using the DeepFX setting hand piece (Ultrapulse, Lumenis), performed under general anaesthetic at 4-6 week intervals. All treatments consisted of a single pass of 300Hz, 5% density and 50mJ energy with minimal overlapping
  Other Names: Ablative Fractional CO2 laser
  Arms: Treatment

SUMMARY:
This study evaluates the effect effect of ablative fractional CO2 laser (AFCO2L) on burns scar appearance and dermal architecture at 6 weeks and up to 3-years post-treatment. Half of the scar will receive AFCO2L and half the scar will receive standard care.

DETAILED DESCRIPTION:
Ablative fractional CO2 laser (AFCO2L) is emerging as a promising scar treatment for burns patients. Fractionated delivery of CO2 laser treatment leaved columns of undamaged skin to quickly re-epithelialize and has reduced the previously higher risk profile of unfractionated ablative laser delivery in terms of permanent pigmentation changes, higher rates of infection and scarring. The exact mechanisms of CO2 laser action are still unclear, but likely involve a combination of macroscopic ablative fenestration, microscopic thermal collagen alteration and molecular profile alterations.

Use of AFCO2L for scar management is increasing amongst burn clinicians; consensus opinion and several large series have demonstrated safe and effective result, however robust randomised controlled evidence for the efficacy of CO2 laser on burns scarring is still lacking.

ELIGIBILITY:
Inclusion Criteria:

* Minimum burn injury scar area of 10x10cm
* Vancouver Scar Scale (VSS) score of >5
* ≥6 months following injury
* Patient age 18+ years

Exclusion Criteria:

* Current pregnancy or lactation
* Patients unable to consent (dementia or another cognitive dysfunction)
* Non-English-speaking patients
* Scars on the face or hand (these anatomical areas were considered to be of significant aesthetic and functional importance and thus excluded from the trial )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2015-01-16 (Actual); Study Completion 2015-07-16 (Actual)

PRIMARY OUTCOMES:
Change in modified Vancouver Scar Scale from baseline at 6 weeks post-final treatment | 6 weeks post final treatment
  The Modified Vancouver Scar Scale requires an assessor to rate the patient's scars in 4 domains, each assigning a score to the scar for different qualities (pliability, height, vascularity and pigmentation) from 0 to 4 in pliability and height; and 0 to 3 in vascularity and pigmentation, where 0 is a 'normal' score as close to normal skin as possible and a score of 3 or 4 would indicate a poor outcome, dissimilar to normal skin. The minimum total score is 0 (very good scar) and maximum score is 14 (very bad scar)
Change in Patient Scar Assessment Scale (patient element of the POSAS scale) from baseline at 6 weeks post-final treatment | 6 weeks post final treatment
  Patient element of the POSAS scale (Patient and Observer Scar Assessment Scale) version 2.0. The scale asks the patient to rate their scars in 6 domains, each assigning a score to the scar for different qualities (pain, itch, colour, stiffness, thickness irregularity and overall opinion) from 1 to 10, where 1 is a very good score and 10 is a very poor score. The minimum total score is 7 (very good scar) and maximum score is 70 (very bad scar)
Change in Scar histology from baseline at 6 weeks post-final treatment | 6 weeks post final treatment
  3mm punch biopsies from treatment and control segments of scar looking at dermal architecture in terms of collagen fibre thickness and orientation

SECONDARY OUTCOMES:
Change in Scar histology from baseline at 48-72 hours after the first treatment | 48-72 hours after the first treatment
  3mm punch biopsies from treatment and control segments of scar looking at dermal architecture in terms of collagen fibre thickness and orientation
Change in modified Vancouver Scar Scale from baseline at 2-3 years post-final treatment | 2-3 years after the final treatment
  The Modified Vancouver Scar Scale requires an assessor to rate the patient's scars in 4 domains, each assigning a score to the scar for different qualities (pliability, height, vascularity and pigmentation) from 0 to 4 in pliability and height; and 0 to 3 in vascularity and pigmentation, where 0 is a 'normal' score as close to normal skin as possible and a score of 3 or 4 would indicate a poor outcome, dissimilar to normal skin. The minimum total score is 0 (very good scar) and maximum score is 14 (very bad scar)
Change in Patient Scar Assessment Scale (patient element of the POSAS scale) from baseline at 6 weeks post-final treatment | 2-3 years after the final treatment
  Patient element of the POSAS scale (Patient and Observer Scar Assessment Scale) version 2.0. The scale asks the patient to rate their scars in 6 domains, each assigning a score to the scar for different qualities (pain, itch, colour, stiffness, thickness irregularity and overall opinion) from 1 to 10, where 1 is a very good score and 10 is a very poor score. The minimum total score is 7 (very good scar) and maximum score is 70 (very bad scar)
Change in Scar histology from baseline at 2-3 years post-final treatment | 2-3 years after the final treatment
  3mm punch biopsies from treatment and control segments of scar looking at dermal architecture in terms of collagen fibre thickness and orientation

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Wood, FRACS, Study Director — UWA and State Burns Unit WA

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months of study completion
Access Criteria: By liaison with principal investigator